CLINICAL TRIAL: NCT00748670
Title: An Open, Prospective, Multicenter Study to Evaluate Treatment of Edentulous Upper Jaws With an Implant-Supported Prosthesis Retained by Astra Tech Dental Implants, Fixture Micro-Macro in Patients With Poor Bone Quality
Brief Title: Treatment With Fixture Microthread™ in Patients With Poor Bone Quality and no Teeth in the Upper Jaw, When Using Two-Stage Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision to modify the product under study as a result of feedback regarding subjective feeling during installation procedure. For more info, see brief summary.
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Head of Therapeutic Area Dental, Clinical Research, Astra Tech AB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YA-MMF-0003
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2008-09-08 (Estimated); Status verified 2008-09

CONDITIONS: Jaw, Edentulous; Poor Bone Quality
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Device: Fixture MicroThread (Micro-Macro)

INTERVENTIONS:
Device: Fixture MicroThread (Micro-Macro) — Fixture MicroThread (Micro-Macro) Ø 3.5 and 4.0 mm in lengths of 9, 11, 13, 15 and 17 mm.

SUMMARY:
The primary objective of the study is to evaluate the long-term survival rate of individual implants and prostheses when treating edentulous upper jaws of poor bone quality with Fixture MicroThread™ (Micro-Macro).

Clinical study recruitment was stopped in year 2000 due to a decision to modify the product under study. This was a result of feedback regarding the subjective feeling during the installation procedure. There were no safety concerns w/r to the study products. Patients already included and treated in the study were monitored for the full duration of the study in accordance with the clinical study protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years of age
* Bone quality class III or IV, (according to Lekholm & Zarb16)
* Willing to give signed informed consent

Exclusion Criteria:

* Need for bone augmentation of the maxilla
* Tobacco smoking more than 5 cigarettes/day
* Any systemic disease or condition that would compromise post-operative healing and/or osseointegration
* Systemic corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
* Unable or unwilling to return for follow-up visits
* Bruxism or other parafunctional activity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 1999-09; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Implant survival | Continuously during 5,5 years after implant placement

CONTACTS AND LOCATIONS:
Overall Officials: Clark Stanford, D.D.S., Ph.D., Principal Investigator — University of Iowa, College of Dentistry, Dow's Institute for Dental Research
Locations (3):
- University of Iowa, College of Dentistry, Dow's Institute for Dental Research, Iowa City, Iowa, United States
- Sweden (2):
  - Specialisttandvården, Avd för Oral Protetik, Länssjukhuset Gävle-Sandviken, Gävle
  - Odontologiska kliniken, Länssjukhuset, Halmstad